CLINICAL TRIAL: NCT00067704
Title: Efficacy of an Emotional Disclosure Intervention in HIV
Brief Title: Emotional Disclosure in HIV
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Miami (Other)
Collaborators: National Center for Complementary and Integrative Health (NCCIH) (NIH)
Responsible Party: Principal Investigator, Gail Ironson, Professor, University of Miami
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 20020511; R01AT002035 (NIH)
Record Dates: First submitted 2003-08-25; First posted 2003-08-27 (Estimated); Last update posted 2015-10-14 (Estimated); Status verified 2015-10

CONDITIONS: HIV Infections
Keywords: Complementary Therapies
MeSH Terms: conditions — HIV Infections

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Trauma writing (Experimental): Four sessions of writing about traumatic experiences.
  Interventions: Behavioral: Trauma writing
- Writing about daily events (Sham Comparator): Four sessions of writing about their daily experiences.
  Interventions: Behavioral: Writing about daily events

INTERVENTIONS:
Behavioral: Trauma writing
  Arms: Trauma writing
Behavioral: Writing about daily events
  Arms: Writing about daily events

SUMMARY:
The specific objective of this study are to examine whether or not a treatment aimed at emotional disclosure may have beneficial psychological, health and immune effects for HIV infected individuals. The goal of the current study is to test the efficacy of emotional disclosure through writing in patients with HIV infection. We will compare emotional disclosure through writing about traumatic experiences (experimental intervention) to a control intervention (writing about emotionally neutral topics). [Note that HIV RNA viral load, CD4 T cells, urinary cortisol, health related dysfunction, psychological distress, and medication adherence are the 6 primary outcome variables.

ELIGIBILITY:
Inclusion Criteria

* 18-65 years of age inclusive
* At least 8 years of formal education
* Literate
* Fluent in English

All of the following three must apply:

* No active Category C HIV AIDS-defining symptoms
* CD4 T-lymphocyte count between 150-499
* Viral load >1000

Exclusion Criteria

* Less than 8 years formal education
* Illiterate or non-English speaking
* Active systemic diseases that would interfere with participation
* Current alcohol or substance dependence
* Planned change in HIV medication in the next 6 months, or recent change in past 2 months
* Introduction of antidepressant medication within 30 days of study start
* Current psychological counseling, cognitive behavior therapy, support group or other psychological therapy, or plans to start any of the above
* Diagnosis of PTSD or major depression
* Unable to attend at least 4 treatment sessions

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 283 (Actual)
Dates: Start 2004-02; Primary Completion 2012-11 (Actual); Study Completion 2012-11 (Actual)

PRIMARY OUTCOMES:
Decrease in psychological distress | 1 year

SECONDARY OUTCOMES:
Increase in CD4 T-lymphocytes | 1 year
Decrease in the number of HIV symptoms | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Gail Ironson, MD, Principal Investigator — University of Miami Dept. of Psychology & Behavioral Medicine
Locations (1):
- University of Miami Dept. of Psychology & Behavioral Medicine, Coral Gables, Florida, United States